CLINICAL TRIAL: NCT06630299
Title: A Phase 3, Randomized, Open-Label, Active-Controlled Study to Evaluate a Switch to an Oral Weekly Islatravir/Lenacapavir Regimen in People With HIV-1 Who Are Virologically Suppressed on Standard of Care
Brief Title: Study to Compare an Oral Weekly Islatravir/Lenacapavir Regimen With Standard of Care in Virologically Suppressed People With HIV-1
Acronym: ISLEND-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-563-5926; 2024-514047-28 (Other: European Medicines Agency)
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: HIV-1-Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ISL/LEN (Experimental): Participants will receive an initial dose of ISL/LEN (Dose A), followed by once weekly ISL/LEN (Dose B) from Day 8 onwards up to Week 96.
  Interventions: Drug: ISL/LEN
- Standard of Care Treatment (Active Comparator): Participants will continue standard of care treatment with 2-3 ARVs up to Week 96:
  * Integrase Strand Transfer Inhibitor (INSTI) class: INSTI combined with 1 or 2 nucleoside reverse transcriptase inhibitors (NRTIs; bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF; coformulated; Biktarvy®), dolutegravir (DTG)/abacavir (ABC)/lamivudine (3TC), DTG+ TAF or TDF (TXF)/emtricitabine (FTC; Emtriva®), DTG/tenofovir disoproxil fumarate (TDF; Viread®)/3TC, DTG/3TC, raltegravir (RAL) + TXF/FTC, RAL+TDF/3TC, elvitegravir (EVG; Vitekta®)/cobicistat (c; Tybost®)/TXF/FTC), or
  * PI class: Boosted protease inhibitor (PI) combined with 2 NRTIs (darunavir/cobicistat/emtricitabine/tenofovir alafenamide (D/C/F/TAF; coformulated), boosted darunavir (DRV)+TXF/FTC, boosted DRV+TDF/3TC), or
  * NNRTI class: Nonnucleoside reverse transcriptase inhibitor (NNRTI) combined with 2 NRTIs (doravirine (DOR)/TDF/3TC, DOR+TXF/FTC, DOR+TDF/3TC, rilpivirine (RPV)/TXF/FTC, RPV+TXF/FTC, RPV+TDF/3TC)
  Interventions: Drug: ISL/LEN; Drug: Antiretroviral Combinations
- Extension Phase (Experimental): At the end of randomized treatment visit, if safety and efficacy of ISL/LEN are demonstrated following review of randomized data, participants will be given the option to receive ISL/LEN tablets in an extension phase until ISL/LEN becomes available or until the sponsor elects to discontinue the study, whichever occurs first.
  Participants receiving ISL/LEN during the randomized phase will continue to take ISL/LEN weekly.
  Participants receiving standard of care during the randomized phase will take an initial dose of ISL/LEN (Dose A), followed by once weekly ISL/LEN (Dose B) from Day 8 onwards.
  Interventions: Drug: ISL/LEN

INTERVENTIONS:
Drug: ISL/LEN — Tablet administered orally
Drug: Antiretroviral Combinations — 2 or 3 antiretrovirals (ARVs) administered as defined by the investigator, according to the prescribing information.
  Arms: Standard of Care Treatment

SUMMARY:
The goal of this clinical study is to learn more about the safety and efficacy of switching to a once weekly tablet of islatravir/lenacapavir (ISL/LEN) regimen versus continuing standard of care treatment in people with human immunodeficiency virus (PWH) who are virologically suppressed (HIV-1 RNA levels < 50 copies/mL) on a stable standard of care regimen for ≥ 6 months prior to screening. The standard of care includes 2 or 3 medicines, antiretroviral agents (ARVs).

The primary objective of the study is to evaluate the efficacy of switching to oral weekly ISL/LEN tablet regimen versus continuing standard of care in virologically suppressed PWH at Week 48.

ELIGIBILITY:
Key Inclusion Criteria:

* HIV-1 RNA < 50 copies/mL for ≥ 6 months before screening, as documented by:

  1. One HIV-1 RNA < 50 copies/mL immediately preceding the 24 weeks period prior to screening.
  2. Within 24 weeks prior to screening, if HIV-1 RNA results are available, all levels must be < 50 copies/mL.
  3. During the 6 to 12 months period prior to screening, transient detectable viremia ≥ 50 copies/mL is acceptable ("blip") as long as it is not confirmed on 2 consecutive visits.
* Plasma HIV-1 RNA levels < 50 copies/mL at screening.
* Are receiving guideline-recommended standard of care treatment such as International Antiviral Society (IAS), Department of Health and Human Services (DHHS), European AIDS Clinical Society (EACS) consisting of 2 or 3 ARVs for ≥ 6 months prior to screening and willing to continue until Day 1. Individuals in Treatment Group 2 must also be willing to continue their standard of care through at least Week 96.
* Individuals assigned female at birth and of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified methods of contraception.

Key Exclusion Criteria:

* Prior virologic failure.
* Prior use of, or exposure to, ISL or LEN.
* Active, serious infections requiring parenteral therapy within 30 days before randomization.
* Active tuberculosis infection.
* Acute hepatitis within 30 days before randomization.
* Hepatitis B virus (HBV) infection, as determined below at the screening visit:

  1. positive HBV surface antigen OR
  2. positive HBV core antibody and negative HBV surface antibody. Note: individuals found to be susceptible to HBV infection (eg negative hepatitis B surface antibody at the screening visit, regardless of prior HBV vaccination history) should be recommended to receive HBV vaccination.
* Active hepatitis C virus (HCV) coinfection, defined as detectable HCV RNA. Note: individuals with prior/inactive HCV infection (defined as undetectable HCV RNA) may be enrolled.
* Any of the following laboratory values at screening:

  1. Creatinine clearance (CLcr) ≤ 30 mL/min according to the Cockcroft-Gault formula
  2. Alanine aminotransferase (ALT) > 5 x upper limit of normal (ULN)
  3. Direct bilirubin > 1.5 x ULN
  4. Platelets < 50,000/μL
  5. Hemoglobin < 8.0 g/dL

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with HIV-1 RNA ≥ 50 copies/mL at Week 48 as Determined by the United States (US) Food and Drug Administration (FDA)-defined Snapshot Algorithm | Week 48

SECONDARY OUTCOMES:
Proportion of Participants with HIV-1 RNA ≥ 50 copies/mL at Week 96 as Determined by the US FDA-defined Snapshot Algorithm | Week 96
Proportion of Participants with HIV-1 RNA < 50 copies/mL at Week 48 as Determined by the US FDA-defined Snapshot Algorithm | Week 48
Proportion of Participants with HIV-1 RNA < 50 copies/mL at Week 96 as Determined by the US FDA-defined Snapshot Algorithm | Week 96
Change from Baseline in clusters of differentiation 4 (CD4) T-Cell Count at Week 48 | Baseline, Week 48
Change from Baseline in CD4 T-Cell Count at Week 96 | Baseline, Week 96
Proportion of Participants Discontinuing ISL/LEN due to Treatment-Emergent Adverse Events (TEAEs) | First dose date up to Week 96

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (100):
- United States (49):
  - University of Alabama at Birmingham(UAB) 1917 Research Clinic, Birmingham, Alabama
  - Pueblo Family Physicians, Phoenix, Arizona
  - Vv-Tmf-5366229, Los Angeles, California
  - Ruane Clinical Research Group, Los Angeles, California
  - BIOS Clinical Research, Palm Springs, California
  - Vivent Health, Denver, Colorado
  - University of Colorado Clinical and Translational Research Center, Denver, Colorado
  - Yale University; School of Medicine; AIDS Program, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Aids Healthcare Foundation - Northpoint, Fort Lauderdale, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - CAN Community Health, Miami Gardens, Florida
  - Orlando Immunology Center, Orlando, Florida
  - AHF Pensacola, Pensacola, Florida
  - CAN Community Health, Sarasota, Florida
  - BayCare Health System, Inc./St. Joseph's Hospital, Tampa, Florida
  - Triple O Research Institute, P.A., West Palm Beach, Florida
  - Metro Infectious Disease Consultants, P.L.L.C., Decatur, Georgia
  - Mercer University, Department of Internal Medicine, Macon, Georgia
  - Chatham County Health Department, Savannah, Georgia
  - Howard Brown Health Center, Chicago, Illinois
  - Indiana CTSI Clinical Research Center, Indianapolis, Indiana
  - Brigham and Womens's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Community Research Initiative of New England d/b/a Community Resource Initiative (CRI), Boston, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Henry Ford Health, Detroit, Michigan
  - Trinity Health Michigan d/b/a Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - ID Care, Hillsborough, New Jersey
  - Saint Michael's Medical Center, Newark, New Jersey
  - AXCES Research Group, LLC, Santa Fe, New Mexico
  - NewYork-Presbyterian Queens, Flushing, New York
  - Northwell Health/Division of Infectious Diseases, Manhasset, New York
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Health System(DUHS), Durham, North Carolina
  - ECU Health Leo Jenkins Cancer Building, Greenville, North Carolina
  - Rosedale Health and Wellness, Huntersville, North Carolina
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Prisma Health Midlands - Clinical Research Unit, Columbia, South Carolina
  - Central Texas Clinical Research, Austin, Texas
  - North Texas Infectious Diseases Consultants, PA, Dallas, Texas
  - AXCES Research Group, LLC, El Paso, Texas
  - Texas Centers for Infectious Disease Associates, Fort Worth, Texas
  - The Crofoot Research Center, INC., Houston, Texas
  - Clinical Alliance for Research& Education - Infectious Diseases, LLC (CARE-ID), Longview, Texas
  - AXCES Research Group, LLC, Salt Lake City, Utah
  - Clinical Alliance for Research& Education - Infectious Diseases, LLC, Annandale, Virginia
  - MultiCare Rockwood Main Clinic, Spokane, Washington
- Argentina (3):
  - Hospital General de Agudos Dr. J.M. Ramos Mejia, Buenos Aires
  - Fundacion Huesped, Buenos Aires
  - Helios Salud S.A., Buenos Aires
- Australia (5):
  - East Sydney Doctors, Darlinghurst, New South Wales
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Taylor Square Private Clinic, Surry Hills, New South Wales
  - Monash Health, Clayton, Victoria
  - Prahran Market Clinic, South Yarra, Victoria
- Germany (4):
  - Dr. Scholten & Schneeweiß GbR, Cologne
  - University Hospital Hannover, Department for Rheumatology and Immunology, Hanover
  - Mannheimer Onkologie Praxis, Mannheim
  - MVZ München am Goetheplatz, MUC Research GmbH, München
- Japan (7):
  - Chiba University Hospital, Chiba
  - National Hospital Organization Nagoya Medical Center, Nagoya
  - University of the Ryukyus Hospital, Okinawa
  - Osaka City General Hospital, Osaka
  - National Hospital Organization Osaka National Hospital, Osaka Fu
  - Tokyo Medical University Hospital, Tokyo
  - Japan Institute for Health Security National Center for Global Health and Medicine, Tokyo
- Netherlands (2):
  - Amsterdam UMC, Iocation AMC, Amsterdam
  - Leiden University Medical Center (LUMC), Leiden
- Poland (2):
  - Samodzielny Publiczny Wojewodzig Szpital Zespolony Poradnia Nabytych Niedoborow Immunologicznych, Szczecin
  - Wroclawskie Centrum Zorowia Samodzielny Publiczn Zaklad Opieki Zdrowotnej Sp Zoo Osrodek Profilaktyczno-Leczniczy Chorob Zakaznych I Terapi Uzaleznien, Wroclaw
- Puerto Rico (2):
  - HOPE Clinical Research, San Juan, PR
  - Maternal Infant Studies Center(CEMI), San Juan
- South Africa (2):
  - Desmond Tutu Health Foundation, Clinical Trials Unit, Cape Town
  - Perinatal HIV Research Unit, Soweto
- Spain (4):
  - Hospital Germans Trias I Pujol, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- Switzerland (3):
  - Inselspital, Freiburgstrasse 20. Bern, Bern
  - Hopitaux Universitaires de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
- Taiwan (5):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - National Taiwan University Hospital, Taipei
  - Taoyuan General Hospital, Taoyuan
- Thailand (6):
  - The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT), Thai Red Cross AIDS Research, Bangkok
  - Siriraj Hospital, Bangkok
  - Chiang Mai University, Chiang Mai
  - Khon Kaen University, Khon Kaen
  - Bamrasnaradura Infectious Disease Institute, Nonthaburi
  - Institute of HIV Research and Innovation (IHRI), Pathumwan
- United Kingdom (6):
  - Clinical Research Facility -University Hospitals Sussex NHS Foundation Trust, Brighton
  - Harrison Wing Research Unit, Southwark Wing, Guy's Hospital (Guy's & St. Thomas' NHS Foundation Trust), Great Maze Pond
  - Grahame Hayton Unit, Ambrose King Centre, Royal London Hospital (Barts Health NHS Trust), London
  - Royal Free Hospital (Royal Free London NHS Foundation Trust), London
  - Caldecot Centre, King's College Hospital (King's College Hospital NHS Foundation Trust), London
  - Mortimer Market Centre (Central and North West London NHS Foundation Trust), London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06630299